CLINICAL TRIAL: NCT04778358
Title: Pilot Trial to Investigate a Higher Dose of Rekovelle in Oocyte Donors
Brief Title: Higher Dose of Rekovelle in Oocyte Donors
Acronym: REKO15
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IVI Madrid (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1901-MAD-013-JG
Record Dates: First submitted 2021-01-28; First posted 2021-03-03 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: IVF
MeSH Terms: interventions — follitropin delta

STUDY DESIGN:
Intervention Model Description: Oocyte donors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OOCYTE DONORS (Experimental): Administration of a higher dose of Rekovelle (follitropin delta) to increase the ovarian response to 17 oocytes (the optimal range being 15 to 25 oocytes) in an oocyte donor population without compromising safety and efficacy.
  Interventions: Drug: Follitropin Delta, Recombinant

INTERVENTIONS:
Drug: Follitropin Delta, Recombinant — 15 µg of follitropin delta will be administered subcutaneously daily

SUMMARY:
Higher numbers of oocytes have not been shown to increase implantation or live newborn rates, but higher numbers of oocytes are likely to be beneficial in certain treatments. These clinical cases where a high ovarian response can be IVF cycles with genetic diagnosis, patients who need more than one pregnancy or, as in our case, oocyte donation. For this reason, and based on previous studies, investigators intend to increase the ovarian response by increasing the dose of follitropin. This clinical trial aims to evaluate high doses of Rekovelle (follitropin delta) to obtain an average of 17 oocytes in a population of oocyte donors, without affecting the health of the patients.

DETAILED DESCRIPTION:
IVF ovarian stimulation cycles has been shown that the individualization of the medication doses provides clinical results comparable to conventional ovarian stimulation regimens, but also it results in greater treatment safety by significantly reducing the percentage of patients with responses extreme ovaries, and cycle cancellations. These studies have been carried out with the premise that an optimal ovarian response results in obtaining 8-14 oocytes per puncture. Although it has also been shown that larger numbers of oocytes do not increase clinical variables such as implantation rates or live newborn per cycle, it is possible that these numbers of oocytes are insufficient in specific circumstances, for example, patients with a desire to have more pregnancy, patients undergoing IVF cycles with PGT-A, or gamete donors. For these reasons, and thanks to the improvements in cryopreservation programs and the induction of oocyte maturation with GnRH agonists, it is necessary to design protocols for the individualization of doses of medication aimed at obtaining greater quantities of oocytes. The objective of this pilot study is the evaluation of higher doses of Rekovelle (follitropin delta) aimed at obtaining 17 oocytes in voluntary donors.

ELIGIBILITY:
Inclusion criteria:

Patients who meet the following inclusion criteria will be candidates to participate in the trial.

* Signed and dated informed consent.
* Oocyte donors between 18 and 35 years of age, both inclusive.
* Presence of at least 6 antral follicles in each ovary on the day of start of stimulation.
* Oocyte donors in their first or second donation cycle.

Exclusion criteria:

Patients who meet the following criteria will not be able to participate in the clinical trial:

* Simultaneous participation in another clinical trial
* Participation in another clinical study before inclusion in this study that could affect its objectives.
* Donors diagnosed with polycystic ovary syndrome according to the Rotterdam criteria (4)
* Endometriosis level III / IV
* Use of hormonal contraceptives (oral or vaginal) in the cycle prior to inclusion.
* Use of Estradiol Valerate for cycle synchronization in the cycle prior to inclusion.
* Family history of hereditary diseases
* Presence of abnormal karyotype
* Positive for any sexually transmitted disease

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Assest the dose of 15µg of follitropin delta aimed at obtaining 17 oocytes (considering the optimal range of oocytes from 15 to 25). | Number of oocytes obtained inmediatly after the ovarian puncture in visit 5
  To evaluate the number of oocytes of a fixed dose of 15µg of the drug Rekovelle (follitropin delta) during the entire stimulation of oocyte donors aimed at obtaining 17 oocytes (considering the optimal range of oocytes from 15 to 25).
Measure the incidence of ovarian hyperstimulation syndrome using15µg of follitropin delta aimed at obtaining 17 oocytes | Through the study completion, an average 1 month.
  Evaluate with a GOLAN scale.
  Golan classification:
  Classify early or late ovarian hyperstimulation syndrome, according to clinic, ultrasound and laboratory tests
  Mild ovarian hyperstimulation:
  * Grade 1 Abdominal discomfort and bloating
  * Grade 2 Grade 1 + nausea, vomiting, or diarrhea. Ovaries enlarged 5-12 cm in ø
  Moderate Hyperstimulation:
  • Grade 3 Grade 2 + ultrasound signs of ascites
  Severe hyperstimulation:
  * Grade 4 Grade 3 + clinical ascites, respiratory distress, hydrothorax
  * Grade 5 Grade 4 and hemoconcentration, hypovolemia, impaired coagulation and renal function (oligo / anuria)

SECONDARY OUTCOMES:
Number of mature oocytes | Number of madure oocytes obtained inmediatly after the puncture in visit 5
  Evaluate the number of mature oocyte
Duration of stimulation in days | Number of days during the ovarian stimulation up to 20 days
  Evaluate the duration of stimulation in days
Number of blasts | 4-6 days after fertilization and before implantation in the endometrium during the treatment.
  Early stage of embryonic development that appears 4-6 days after fertilization and before implantation in the endometrium
Blast quality | 4-6 days after fertilization and before implantation in the endometrium during the treatment.
  Blast quality according to the Gardner scale, classification of blastocysts, where in addition to the structure of the inner cell mass (ICM) and cells of the trophectoderm, it provides a degree of expansion
Degree of satisfaction with the infertility treatment | At the end of the treatment, an average 1 month.
  Degree of satisfaction with the infertility treatment according to the EFESO, Questionnaire designed to know the degree of satisfaction of women who undergo ovarian stimulation treatment to treat their infertility questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Valenciano de Infertilidad, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No